CLINICAL TRIAL: NCT04105699
Title: A Multicenter, Prospective, Biomarker-result-blinded Observational Study Evaluating Immunoassay Measurements of Pancreatic Stone Protein Performed on Abionic's abioSCOPE® Device With the PSP Assay on ICU Patients at Risk of Sepsis as an Aid in Identifying Sepsis
Brief Title: Evaluation of Immunoassay Measurements of Pancreatic Stone Protein Performed on abioSCOPE® Device With the PSP Assay on ICU Patients at Risk of Sepsis as an Aid in Identifying Sepsis
Status: Completed | Type: Observational
Sponsor: Abionic SA (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-PSP-002
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Sepsis
Keywords: Sepsis; Pancreatic Stone Protein; Point-of-care device; Immunoassay; Intensive care unit; Abionic
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous serum retained for future investigation related to sepsis biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Device: Blood sampling
  Interventions: Device: Blood sampling

INTERVENTIONS:
Device: Blood sampling — Daily blood sample which will be taken for the PSP measurement using the abioSCOPE as well as another daily sample taken for central analysis of biomarkers of inflammation, infection and/or sepsis (including but not limited to C-reactive protein [CRP] and Procalcitonin [PCT]).

SUMMARY:
This is a multicenter, prospective, biomarker-result-blinded observational study evaluating immunoassay measurements of pancreatic stone protein (PSP) performed on Abionic's abioSCOPE device with the PSP assay on ICU patients at risk of sepsis as an aid in identifying sepsis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision and understanding of signed and dated written informed consent by patient or legally designated representative prior to any mandatory study-specific procedures, sample collection, or analysis.
* 2. Male or female, aged ≥ 18 years.
* 3. Admitted to ICU on the day of screening, with expectation that patient will require ICU management for a minimum of 24 hours.

Exclusion Criteria:

* 1. Expected to die within 24 hours no matter what therapy is given, from the time of screening.
* 2. Suffering on ICU admission or study entry from or known acute or chronic pancreatitis or pancreatic cancer).
* 3. Admitted to ICU due to elective cardiac surgery with an uncomplicated stay anticipated.
* 4. Patients having a valid Do Not Resuscitate order.
* 5. Previous ICU admission during this hospital stay
* 6. Confirmed COVID-19 as reason for ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU admitted patients at risk of developing sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 544 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Ability of the abioSCOPE PSP assay performed on day 1 of a participant's ICU admission to correctly identify those with sepsis. | Day 1
  Assess the clinical sensitivity and specificity of the abioSCOPE PSP assay obtained on day 1 of ICU stay to identify sepsis within 3 days, based on EIRC assessment of sepsis.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Mercy Health St. Vincent, Toledo, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Undecided